CLINICAL TRIAL: NCT01628354
Title: A Study to Investigate the Safety and Efficacy of Lucentis (Ranibizumab) in Patients With CNV Due to Causes Other Than AMD and in Patients Where Pigment Epithelial Detachments Are the Primary Manifestation of Their AMD.
Brief Title: Study to Investigate the Safety and Efficacy of Ranibizumab in Patients With Choroidal Neovascularisation Due to Causes Other Than Age Related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Robyn Guymer, Professor Robyn Guymer, Head Macular Research Unit, Department of Ophthalmology., University of Melbourne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHG
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Choroidal Neovascularization; Retinal Pigment Epithelial Detachment
Keywords: Choroidal neovascularization; Lucentis
MeSH Terms: conditions — Choroidal Neovascularization; Retinal Detachment | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ranibizumab — All patients will receive an intravitreal injection of ranibizumab 0.5 mg at baseline (visit 1; month 0) then a subsequent intravitreal injection at month 1 (visit 2) and month 2 (Visit 3). Patients will be reviewed every month thereafter for 12 months at which time it will be determined whether the patient requires retreatment with ranibizumab 0.5 mg based on measurements of visual acuity, Optical coherene tomography (OCT) findings and clinical appearance. A drop of vision of >5 letters or increase in retinal thickness of >100 um on OCT will trigger re-treatment as long as 14 days has elapsed since last treatment.
  Other Names: Lucentis

SUMMARY:
The investigators hypothesize that it is safe and effective to treat patients with choroidal neovascularisation (abnormal blood vessels growing under the retina) secondary to causes other than age related macular degeneration (AMD) and pigment epithelial detachments (blisters of fluid under the retina) secondary to AMD with ranibizumab (Lucentis).

These groups of patients have to date been excluded from the multicentre trials demonstrating significant benefit of Ranibizumab in the treatment of AMD.

DETAILED DESCRIPTION:
Hypothesis

1. That it is safe to treat patients with choroidal neovascularisation (CNV) secondary to causes other than age related macular degeneration (AMD) with ranibizumab
2. That treatment of CNV secondary to causes other than AMD with ranibizumab is effective
3. That treatment of pigment epithelial detachments (PEDs) secondary to CNV from AMD with ranibizumab is safe
4. That treatment of pigment epithelial detachments (PEDs) secondary to CNV from AMD with ranibizumab is effective

Objectives

The primary objectives of this study are:

* to investigate the medium term safety and efficacy of Ranibizumab in the treatment of CNV secondary to causes other than AMD (eg. angioid streaks, pseudoxanthoma elasticum, trauma, macular dystrophies, ocular inflammation/choroiditis and idiopathic causes).
* to investigate the medium term safety and efficacy of Ranibizumab in the treatment of PEDs that are secondary to CNV from AMD

These groups of patients have to date been excluded from the multicentre trials demonstrating significant benefit of Ranibizumab in the treatment of AMD.

Strategic goal

To explore the safety and efficacy of intravitreal ranibizumab in patients with CNV due to causes other than AMD for which there is currently no approved or suitable treatment. Our goal is also to explore the safety and efficacy of intravitreal ranibizumab in patients where PEDs have been the primary manifestation of he CNVM secondary to AMD.

To use a treatment protocol in which the frequency of intraocular injection is minimised.

Background

Although the stimuli that induce choroidal neovascularisation (CNV) are unknown, there is evidence suggesting that angiogenic factors such as vascular endothelial growth factor (VEGF) and basic fibroblast growth factor play a role in the pathogenesis of CNV. VEGF is a polypeptide secreted by the retinal pigmented epithelium that exerts a potent proliferative effect specifically on vascular endothelial cells. The presence of supernormal amounts of VEGF in surgically excised human CNV provides evidence that VEGF contributes to CNV lesion formation in AMD and also in CNV due to other causes. In CNV, the newly formed vessels have a tendency to leak blood and fluid, causing symptoms of scotoma and metamorphopsia. The new vessels are accompanied by proliferation of fibrous tissue. This complex of new vessels and fibrous tissue can destroy photoreceptors within 3 to 24 months. At the same time that CNV is destroying retinal tissue where it has formed, the lesion can continue to grow throughout the macula, resulting in progressive, severe and irreversible vision loss. Without treatment, most affected eyes will have poor central vision within 2 years.

Ranibizumab is an anti-VEGF antibody fragment that blocks VEGF activity in patients with neovascular AMD. Its mechanism of action involves forming a complex with VEGF thereby preventing it from binding to its receptors. It is derived from a 149kDa parent murine monoclonal anti¬VEGF antibody and consists solely of a 48 kDa single antigen¬binding portion of that monoclonal antibody without the constant region; thus ranibizumab is approximately one-third the size of the full-length antibody. With this reduced size, ranibizumab is able to penetrate more efficiently through the many retinal cell layers following intravitreal injection as compared with a full¬length MAb (Mordenti et al, 1999).

More than 900 patients have been treated with ranibizumabin clinicla trials to date. It is now registered for use in the USa and is available in Australia under a special access scheme. Results have shown that ranibizumab is safe and well tolerated. Common ocular side effects were mild to moderate and included conjunctival hemorrhage, eye pain and vitreous floaters. Serious ocular adverse events were uncommon (<1%) and included uveitis and endophthalmitis. No discernible patterns of change in circulating levels of VEGF have been observed. In multiple dose studies, the majority of patients experienced little or no change in intraocular pressure (lOP) after treatment. Efficacy in the treatment of CNV secondary to AMD has also been demonstrated in several studies. In a recent phase III study, approximately 95% of patients treated with ranibizumab avoided moderate vision loss compared to 62% in the sham-controlled group while 71-75% maintained or improved vision compared to 29% in the sham-controlled group at 12 months. Vision improved by more than 15 letters in 25% of patients treated with 0.3 mg of ranibizumab and 34% of patients treated with 0.5 mg of ranibizumab compared to 5% of patients in the sham-controlled group. This treatment benefit observed at 12 months was maintained out to 24 months.

Subretinal choroidal neovascularisation (CNV) can occur due to other conditions other than AMD such as pseudoxanthoma elasticum, trauma, macular dystrophies and choroiditis (inflammation of the choroid). Often, patients with CNV due to conditions other than AMD such as those mentioned are relatively young compared to those without AMD, and have a much greater chance of retaining good vision if the CNV can be controlled. Currently, the only treatments available for these patient groups are photodynamic therapy (PDT) with Visudyne or conventional laser therapy. Neither of these treatments however, offer much hope of improving vision. Our experience of using PDT with Visudyne in these individuals is that, relative to those patients with AMD, these non AMD treatments need far fewer treatments and that their final visual acuity is much greater. Given that CNV secondary to other causes does respond to PDT, we extrapolate that these CNV will respond to the new generation of anti-vascular endothelial growth factor (VEGF) agents such as Ranibizumab that have been shown to be effective in the treatment of CNV secondary to AMD.

To date, all of the multicentre trials with ranibizumab have excluded these non AMD patients thus limiting their access to the new generation of intravitreal anti - VEGF treatments.

CNV secondary to AMD can result in pigment epithelial detachments (PEDs) that can lead to the same devastating loss of vision. PEDs have always been difficult to treat, often because they rip as a result of any treatment such as PDT or laser. To date there is no proven treatment for this relatively common presentation of CNV secondary to AMD. They have always been excluded from the multi-centred international studies with Ranibizumab because the active area of CNV did not make up more than 50% of the lesion. This is because the pigment epithelial detachment is considered part of the lesion but is not considered an active part of the lesion. As such very little information is known about the potential for effective treatment with the new generation of anti VEGF drugs.

There have been case reports of resolution of PEDs and improvement of vision after treatment with Bevacizumab (derived from the same parent molecule as ranibizumab) that has been used in an off label setting for the treatment of wet AMD. We believe that these PEDs will similarly respond to treatment with ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with choroidal neovascular membrane secondary to causes other than AMD or patients with Pigment epithelial detachments secondary to AMD where there is demonstrated progression of the disease.
* Total lesion area < 12 disc areas.
* Total area of CNV within the lesion must be > 50% of total lesion area in the first category of recruits, but not in those with PEDs.
* Best corrected visual acuity of 20/40 to 20/320 in the study eye.
* Willing and able to give informed consent

Exclusion Criteria:

* Prior treatment in the study eye with, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy or other anti VEGF treatments.
* History of submacular surgery or other surgical intervention in the study eye, glaucoma filtration surgery, corneal transplant surgery,
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within one month preceding baseline,
* Extracapsular extraction of cataract with phacoemulsification within three months preceding baseline, or a history of post-operative complications within the last 12 months preceding baseline in the study eye (uveitis, cyclitis, etc.),
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication),
* Aphakia with absence of the posterior capsule in the study eye,
* Active intraocular inflammation (grade trace or above) in the study eye,
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis, as well as idiopathic or autoimmune-associated uveitis in either eye,
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye,
* Presence of a retinal pigment epithelial tear involving the macula in the study eye,
* Subfoveal fibrosis or atrophy in the study eye.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity | 12 months

SECONDARY OUTCOMES:
Mean change from baseline in retinal thickness | 12 months
Mean number of ranibizumab injections required over 12 months | 12 months
Ocular and systemic adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robyn H Guymer, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Royal Victorian Eye and Ear Hospital, Melbourne, Victoria, Australia